CLINICAL TRIAL: NCT01691313
Title: Randomized, Double-blind, Placebo-controlled Dose Modification Study to Evaluate the Safety and Efficacy of Single Doses of Vanoxerine for Conversion of Subjects With Recent Onset Atrial Fibrillation or Flutter to Normal Sinus Rhythm
Brief Title: Safety and Efficacy of Vanoxerine for Conversion of Atrial Fibrillation or Flutter to Normal Sinus Rhythm
Acronym: COR-ART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laguna Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRX-VN-002
Record Dates: First submitted 2012-09-20; First posted 2012-09-24 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-11

CONDITIONS: Symptomatic Atrial Fibrillation; Atrial Flutter
Keywords: vanoxerine; atrial fibrillation; atrial flutter; a-fib
MeSH Terms: conditions — Atrial Flutter; Atrial Fibrillation | interventions — vanoxerine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- vanoxerine 200mg (Experimental): vanoxerine HCl 200mg single dose (2x 100 mg oral capsule)
  Interventions: Drug: Vanoxerine
- placebo (Placebo Comparator): placebo to match vanoxerine oral capsule
  Interventions: Drug: Placebo
- vanoxerine 300mg (Experimental): vanoxerine HCl 300 mg single dose (3x 100mg oral capsules)
  Interventions: Drug: Vanoxerine
- vanoxerine 400mg (Experimental): vanoxerine HCl 400 mg single dose (4x 100 mg oral capsules)
  Interventions: Drug: Vanoxerine

INTERVENTIONS:
Drug: Vanoxerine — single oral dose
  Other Names: GBR12909
  Arms: vanoxerine 200mg; vanoxerine 300mg; vanoxerine 400mg
Drug: Placebo — single oral dose
  Other Names: Placebo to match vanoxerine
  Arms: placebo

SUMMARY:
Evaluate the safety and efficacy of a single oral dose of vanoxerine compared to placebo, in a dose modification manner, on the conversion of symptomatic atrial fibrillation (a-fib) or flutter of recent onset to normal sinus rhythm.

DETAILED DESCRIPTION:
Vanoxerine has important antiarrhythmic properties and may prove effective in converting AF/AFL to sinus rhythm in subjects with a history of AF. This is a prospective, randomized, double-blinded, placebo-controlled, dose-modifying study in subjects who have been in symptomatic AF or AFL for more than 3 hours and less than 7 days as dated by symptoms, who have AF/AFL documented on ECG at the time of study drug administration, and who satisfy the inclusion and exclusion criteria. The primary objectives of the trial are to evaluate the safety and efficacy of a single oral dose of vanoxerine compared to placebo following oral administration.

ELIGIBILITY:
Inclusion Criteria:

* provide written informed consent,
* male or female 18 years of age or greater; women of child bearing potential must use adequate contraception
* symptomatic AF/AFL for more than 3 hours and less than 7 days (168 hours), as dated by symptoms
* AF/AFL documented by ECG at the start of study drug administration

Exclusion Criteria:

* Systolic blood pressure <100 mmHg.
* Average heart rate <50 bpm.
* Average QTcF (Fridericia correction) >440 ms.
* Average QRS interval >140 ms.
* Paced atrial or ventricular rhythm on ECG.
* Serum potassium <3.5 meq/L (may be corrected prior to randomization).
* Received another intravenous Class I or Class III antiarrhythmic drug within prior 3 days.
* received amiodarone (oral or IV) in prior 3 months.
* Clinical evidence or history of acute coronary syndrome within 30 days prior to randomization.
* Aortic stenosis with aortic valve area equal to or less than 1.0 cm2.
* Rheumatic mitral stenosis with valve area of <1.5 cm2.
* Untreated hyperthyroidism.
* Acute pericarditis.
* AF/AFL as a result of surgery within the last 7 days
* History of failed electrical cardioversion
* History of polymorphic ventricular tachycardia (PVT, e.g. torsades de pointes).
* History or family history of long QT syndrome.
* History of ventricular tachycardia requiring drug or device therapy.
* History of NYHA Heart Failure Class 3 or 4 or recent (within 1 month) onset of heart failure not related to rapid ventricular response AF.
* Ejection fraction (EF) of 35% or less.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard C Dittrich, MD, Study Director — ChanRx Corp.
Locations (6):
- Israel (4):
  - Ashkelon
  - Haifa
  - Nazareth
  - Safed
- Russia (2):
  - Moscow
  - Saint Petersburg

REFERENCES:
- [Result] Dittrich HC, Feld GK, Bahnson TD, Camm AJ, Golitsyn S, Katz A, Koontz JI, Kowey PR, Waldo AL, Brown AM. COR-ART: A multicenter, randomized, double-blind, placebo-controlled dose-ranging study to evaluate single oral doses of vanoxerine for conversion of recent-onset atrial fibrillation or flutter to normal sinus rhythm. Heart Rhythm. 2015 Jun;12(6):1105-12. doi: 10.1016/j.hrthm.2015.02.014. Epub 2015 Feb 12. PMID 25684233

RESULTS

PARTICIPANT FLOW:
Groups:
- Vanoxerine 200mg: vanoxerine 200 mg (2x 100mg oral capsules)
  Vanoxerine: single oral dose
- Vanoxerine 300mg: vanoxerine 300 mg (3x 100 mg oral capsules) single oral dose
- Vanoxerine 400mg: vanoxerine 400 mg (4x100mg oral capsules) single oral dose
Period: Overall Study
Arm/Group | Vanoxerine 200mg | Placebo | Vanoxerine 300mg | Vanoxerine 400mg
Started | 22 | 32 | 25 | 25
Completed | 22 | 32 | 25 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vanoxerine 200mg: vanoxerine oral capsule, 200mg
  Vanoxerine: single oral dose
- Vanoxerine 300mg: vanoxerine oral capsule, 300mg
  Vanoxerine: single oral dose
- Vanoxerine 400mg: vanoxerine oral capsule, 400mg
  Vanoxerine: single oral dose
- Total: Total of all reporting groups
Arm/Group | Placebo | Vanoxerine 200mg | Vanoxerine 300mg | Vanoxerine 400mg | Total
Number analyzed (Participants) | 32 | 22 | 25 | 25 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (12.2) | 61.7 (12.2) | 63.4 (9.4) | 68.4 (9.6) | 64 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 9 | 13 | 41
  Male | 22 | 13 | 16 | 12 | 63

OUTCOME MEASURES:

1. Primary Outcome: Conversion to Sinus Rhythm
Description: proportion of subjects who convert to sinus rhythm through 4 hours after start of study drug
Time Frame: baseline through 4 hours
Measure: Number; unit: participants
Arm/Group | Placebo | Vanoxerine 200mg | Vanoxerine 300mg | Vanoxerine 400mg
Number analyzed (Participants) | 32 | 22 | 25 | 25
participants | 4 | 4 | 11 | 13

2. Primary Outcome: Conversion to Sinus Rhythm
Description: proportion of subjects who convert to sinus rhythm through 24 hours after start of study drug
Time Frame: baseline through 24 hours
Measure: Number; unit: participants
Arm/Group | Placebo | Vanoxerine 200mg | Vanoxerine 300mg | Vanoxerine 400mg
Number analyzed (Participants) | 32 | 22 | 25 | 25
participants | 10 | 13 | 16 | 21

ADVERSE EVENTS:
Arm/Group | Placebo | Vanoxerine 200mg | Vanoxerine 300mg | Vanoxerine 400mg
Serious Adverse Events (participants affected / at risk) | 0/32 | 1/22 | 1/25 | 0/25
Other Adverse Events (participants affected / at risk) | 3/32 | 3/22 | 8/25 | 17/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=32) | Vanoxerine 200mg (N=22) | Vanoxerine 300mg (N=25) | Vanoxerine 400mg (N=25)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=32) | Vanoxerine 200mg (N=22) | Vanoxerine 300mg (N=25) | Vanoxerine 400mg (N=25)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
ECG QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalized ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other